CLINICAL TRIAL: NCT01600599
Title: Efficacy in Controlling Bleeding Post-coronary Bypass Surgery Using Combination of Local Application of Tranexamic Acid and Intravenous Tranexamic Compared to Intravenous Tranexamic Acid Alone. A Randomized Controlled Trial
Brief Title: Reducing Post Operative Bleeding Following Cabg
Acronym: LATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Theevashini Krishnasamy, MBChB, MRCS, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 180880
Record Dates: First submitted 2012-05-02; First posted 2012-05-17 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Post CABG Bleeding
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV & topical TA (Active Comparator): patients in this group will receive both intravenous & topical tranexamic acid
  Interventions: Drug: Tranexamic Acid
- IV tranexamic acid & Topical Saline (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Tranexamic Acid — intravenous 1g and topical 1g
  Arms: IV & topical TA
Drug: saline — 100mls of topical saline
  Arms: IV tranexamic acid & Topical Saline

SUMMARY:
The purpose of this study is to assess the efficacy of IV Tranexamic Acid and topical Tranexamic Acid to control post op bleeding following Coronary Artery Bypass Graft Surgery using Cardiopulmonary Bypass.

DETAILED DESCRIPTION:
Coagulopathy is a common problem after open heart surgery using cardiopulmonary bypass (CPB). Some bleeding is significant enough to require early re-exploration to control hemorrhage in 2-4% of patients.(1,2) In adults, excessive post-operative bleeding occurs in association with repeat operations, emergency procedures, female gender, small body mass index, older age, peripheral vascular disease, renal insufficiency ( creatinine > 1.8g/dL) , poor nutrition ( albumin < 4g/dL) and in patients who have experienced prolonged CPB durations. (3,4)

Factors that contribute to coagulopathy after coronary artery bypass grafting (CABG) using CPB include thrombocytopenia, acquired platlet dysfunction, loss of clotting factors, free heparin and increased fibrinolysis. (5-7). Lemmer and Colleagues (8) found that extracorporeal circulation results in significant fibrinolysis, as reflected by increased concentrations of plasmin and fibrin degradation products (FDP), both of which have deleterious effects on platlet function. Fibrinolysis was found to be responsible for 25-45% of significant post-bypass bleeding. (9)

Many antifibrinolytic agents have been used to reduce post-bypass bleeding. These include ε- Aminocaproic Acid (10), Aprotinin (11) and Tranexamic Acid (TA) (12).

TA has been found to bind to lysine binding sites of plasmin and plasminogen. Saturation of these sites displaces plasminogen from the fibrin surface thus inhibiting fibrinolysis.(13). TA has been used both systemically and topically.

Due to the natural barrier properties of the pericardium, which prevents the free diffusion of substances, experimental studies have shown that the local application of different medications in to the pericardial cavity can lead to desirable therapeutic effects without significant systemic absorption. (14-16)

There has been a systemic review and meta-analysis study done looking at 8 trials (622 patients) using topical antifibrinolytic agents (aprotinin and tranexamic acid). No adverse effects were reported following usage of topical antifibrinolytics.(17)

Topical TA has also been successfully used in controlling bleeding in bladder, gynaecological, oral, & oropharyngeal surgeries. (18-20)

There has been no authors thus far who have compared application of intravenous TA to combination of application of intravenous TA and topical TA.

This study is based on a hypothesis that the combination of intravenous (IV) TA and topical TA administration will significantly reduce the amount of post-op bleeding significantly following CABG using CPB.

ELIGIBILITY:
Inclusion Criteria:

* primary isolated CABG

Exclusion Criteria:

* patients who will have combined procedure
* redo-surgery
* bleeding diathesis (Haemophilia or platelet count ,100 x 109 L1)
* renal impairment (Creatinine > 130umol/L)
* known allergy to TA
* recent (< 7 days before surgery) intake of anti-platelets (eg Aspirin, Clopidogrel, Ticlid) or heparin administration within 48 hours of operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
chest drain output | 4 days
  chest drain output (in mls) following post CABG in the 1st hour and total drain output when the drain is removed.

CONTACTS AND LOCATIONS:
Overall Officials: theevashini krishnasamy, MBChB, MRCS, Principal Investigator — University of Malaya
Locations (1):
- Pusat Perubatan University Malaya, Petaling Jaya, Selangor, Malaysia

REFERENCES:
- [Background] Munoz JJ, Birkmeyer NJ, Dacey LJ, Birkmeyer JD, Charlesworth DC, Johnson ER, Lahey SJ, Norotsky M, Quinn RD, Westbrook BM, O'Connor GT. Trends in rates of reexploration for hemorrhage after coronary artery bypass surgery. Northern New England Cardiovascular Disease Study Group. Ann Thorac Surg. 1999 Oct;68(4):1321-5. doi: 10.1016/s0003-4975(99)00728-6. PMID 10543500
- [Background] Moulton MJ, Creswell LL, Mackey ME, Cox JL, Rosenbloom M. Reexploration for bleeding is a risk factor for adverse outcomes after cardiac operations. J Thorac Cardiovasc Surg. 1996 May;111(5):1037-46. doi: 10.1016/s0022-5223(96)70380-x. PMID 8622301
- [Background] Magovern JA, Sakert T, Benckart DH, Burkholder JA, Liebler GA, Magovern GJ Sr, Magovern GJ Jr. A model for predicting transfusion after coronary artery bypass grafting. Ann Thorac Surg. 1996 Jan;61(1):27-32. doi: 10.1016/0003-4975(95)00808-X. PMID 8561579
- [Background] Despotis GJ, Filos KS, Zoys TN, Hogue CW Jr, Spitznagel E, Lappas DG. Factors associated with excessive postoperative blood loss and hemostatic transfusion requirements: a multivariate analysis in cardiac surgical patients. Anesth Analg. 1996 Jan;82(1):13-21. doi: 10.1097/00000539-199601000-00004. PMID 8712388
- [Background] Kucuk O, Kwaan HC, Frederickson J, Wade L, Green D. Increased fibrinolytic activity in patients undergoing cardiopulmonary bypass operation. Am J Hematol. 1986 Nov;23(3):223-9. doi: 10.1002/ajh.2830230306. PMID 3766524
- [Background] Harker LA, Malpass TW, Branson HE, Hessel EA 2nd, Slichter SJ. Mechanism of abnormal bleeding in patients undergoing cardiopulmonary bypass: acquired transient platelet dysfunction associated with selective alpha-granule release. Blood. 1980 Nov;56(5):824-34. No abstract available. PMID 6448643
- [Background] Despotis GJ, Santoro SA, Spitznagel E, Kater KM, Cox JL, Barnes P, Lappas DG. Prospective evaluation and clinical utility of on-site monitoring of coagulation in patients undergoing cardiac operation. J Thorac Cardiovasc Surg. 1994 Jan;107(1):271-9. PMID 8283896
- [Background] Lemmer JH Jr, Stanford W, Bonney SL, Breen JF, Chomka EV, Eldredge WJ, Holt WW, Karp RB, Laub GW, Lipton MJ, et al. Aprotinin for coronary bypass operations: efficacy, safety, and influence on early saphenous vein graft patency. A multicenter, randomized, double-blind, placebo-controlled study. J Thorac Cardiovasc Surg. 1994 Feb;107(2):543-51; discussion 551-3. PMID 7508070
- [Background] Kevy SV, Glickman RM, Bernhard WF, Diamond LK, Gross RE. The pathogenesis and control of the hemorrhagic defect in open heart surgery. Surg Gynecol Obstet. 1966 Aug;123(2):313-8. No abstract available. PMID 5913482
- [Background] Daily PO, Lamphere JA, Dembitsky WP, Adamson RM, Dans NF. Effect of prophylactic epsilon-aminocaproic acid on blood loss and transfusion requirements in patients undergoing first-time coronary artery bypass grafting. A randomized, prospective, double-blind study. J Thorac Cardiovasc Surg. 1994 Jul;108(1):99-106; discussion 106-8. PMID 8028387
- [Background] Cosgrove DM 3rd, Heric B, Lytle BW, Taylor PC, Novoa R, Golding LA, Stewart RW, McCarthy PM, Loop FD. Aprotinin therapy for reoperative myocardial revascularization: a placebo-controlled study. Ann Thorac Surg. 1992 Dec;54(6):1031-6; discussion 1036-8. doi: 10.1016/0003-4975(92)90066-d. PMID 1280411
- [Background] Longstaff C. Studies on the mechanisms of action of aprotinin and tranexamic acid as plasmin inhibitors and antifibrinolytic agents. Blood Coagul Fibrinolysis. 1994 Aug;5(4):537-42. PMID 7531000
- [Background] Baek SH, Hrabie JA, Keefer LK, Hou D, Fineberg N, Rhoades R, March KL. Augmentation of intrapericardial nitric oxide level by a prolonged-release nitric oxide donor reduces luminal narrowing after porcine coronary angioplasty. Circulation. 2002 Jun 11;105(23):2779-84. doi: 10.1161/01.cir.0000017432.19415.3e. PMID 12057994
- [Background] Kolettis TM, Kazakos N, Katsouras CS, Niokou D, Pappa L, Koulouras V, Stefanou P, Seferiadis C, Malamou-Mitsi V, Michalis LK, Marselos M, Sideris DA. Intrapericardial drug delivery: pharmacologic properties and long-term safety in swine. Int J Cardiol. 2005 Mar 30;99(3):415-21. doi: 10.1016/j.ijcard.2004.03.004. PMID 15771922
- [Background] Waxman S, Pulerwitz TC, Rowe KA, Quist WC, Verrier RL. Preclinical safety testing of percutaneous transatrial access to the normal pericardial space for local cardiac drug delivery and diagnostic sampling. Catheter Cardiovasc Interv. 2000 Apr;49(4):472-7. doi: 10.1002/(sici)1522-726x(200004)49:43.0.co;2-y. PMID 10751782
- [Background] Abrishami A, Chung F, Wong J. Topical application of antifibrinolytic drugs for on-pump cardiac surgery: a systematic review and meta-analysis. Can J Anaesth. 2009 Mar;56(3):202-12. doi: 10.1007/s12630-008-9038-x. Epub 2009 Feb 12. PMID 19247741
- [Background] Verstraete M. Clinical application of inhibitors of fibrinolysis. Drugs. 1985 Mar;29(3):236-61. doi: 10.2165/00003495-198529030-00003. PMID 2580684
- [Background] Valsecchi A. [Further notes on the topical use of tranexamic acid in the treatment of gynecological hemorrhage]. Minerva Ginecol. 1980 Sep;32(9):825-30. No abstract available. Italian. PMID 7219835
- [Background] Sindet-Pedersen S, Ramstrom G, Bernvil S, Blomback M. Hemostatic effect of tranexamic acid mouthwash in anticoagulant-treated patients undergoing oral surgery. N Engl J Med. 1989 Mar 30;320(13):840-3. doi: 10.1056/NEJM198903303201305. PMID 2648144
- [Background] Abul-Azm A, Abdullah KM. Effect of topical tranexamic acid in open heart surgery. Eur J Anaesthesiol. 2006 May;23(5):380-4. doi: 10.1017/S0265021505001894. Epub 2006 Jan 27. PMID 16438759
- [Background] De Bonis M, Cavaliere F, Alessandrini F, Lapenna E, Santarelli F, Moscato U, Schiavello R, Possati GF. Topical use of tranexamic acid in coronary artery bypass operations: a double-blind, prospective, randomized, placebo-controlled study. J Thorac Cardiovasc Surg. 2000 Mar;119(3):575-80. doi: 10.1016/s0022-5223(00)70139-5. PMID 10694619